CLINICAL TRIAL: NCT04253873
Title: Clinical Study of Apatinib Combined With Temozolomide in the Treatment of Uncontrolled or Repeated High-grade Gliomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: WuHui (Other Government)
Responsible Party: Sponsor-Investigator, WuHui, Doctor, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-AHN02
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: High-grade Gliomas
MeSH Terms: interventions — apatinib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib mesylate + temozolomide (Experimental): Apatinib mesylate tablets (0-14 days, 500 mg, qd), one week apart, then temozolomide (150mg/m2, 5 days);Every 28 days is a cycle, the drug until the disease progress, the toxicity of intolerable.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib mesylate (0-14 days, 500 mg, qd), taken half an hour after a meal (the daily dose should be as much as possible), one week apart, and then given temozolomide (150mg/m2 for 5 Days); every 28 days is a cycle, medication to disease progression, intolerable toxicity, etc.
  Other Names: temozolomide

SUMMARY:
Gliomas are the most common malignant tumors of the central nervous system and are highly invasive. Gliomas account for one-third of central nervous system tumors in adults and children. Interstitial astrocytomas and glioblastomas are also called high-grade gliomas, accounting for 77.5% of all gliomas.

DETAILED DESCRIPTION:
Temozolomide combined with concurrent radiotherapy, followed by 6 cycles of temozolomide adjuvant chemotherapy, can prolong the patient's survival, and the 2-year survival rate has increased from 10.4% to 26.5%. Great progress has been made, but the prognosis for glioma patients remains poor. For patients with poor-quality high-grade gliomas, more effective new treatments are urgently needed to achieve the purpose of survival benefit.

Targeting VEGFs to inhibit tumor angiogenesis has shown good efficacy in a variety of tumors including colon cancer, gastric cancer, lung cancer, liver cancer and breast cancer. However, for gliomas, anti-tumor angiogenesis drugs can improve patient OS Evidence related to PFS is still scarce. Compared with other targeted drugs with multiple kinase targets, apatinib has not only an advantage in price but also less side effects. Therefore, based on relevant data from previous studies, a basic and clinical study of this apatinib combined with temozolomide for high-grade gliomas was performed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 ~ 70 years old, male or female; 2. ECOG score: 0-2 points; 3. Expected survival time ≥ 3 months; 4. Patients diagnosed with high-grade (WHO III, IV) gliomas by pathology, and patients whose disease recurrence is judged by contrast imaging, have at least one measurable lesion on the skull magnetic resonance; 5. Patients who have not been controlled or relapsed after previous first-line standard treatment; 6. The main organs function normally, that is, they meet the following standards:

  1. The blood routine examination standards must be met (no blood transfusion and blood products within 14 days, no correction using G-CSF and other hematopoietic stimulating factors)

     1. HB≥90 g / L;
     2. ANC≥1.5 × 109 / L;
     3. PLT≥80 × 109 / L;
  2. Biochemical inspection must meet the following standards:

     1. TBIL <1.5ULN;
     2. ALT and AST <2.5ULN, but <5ULN for patients with liver metastases;
     3. Serum Cr≤1.25ULN or endogenous creatinine clearance rate> 45 ml / min (Cockcroft-Gault formula); 7. Women of childbearing age must have taken reliable contraceptive measures or performed a pregnancy test (serum or urine) within 7 days before enrollment, with negative results, and be willing to use appropriate methods during the test and 8 weeks after the last dose contraception. For men, consent must be given to appropriate contraception or surgical sterilization during the trial and 8 weeks after the last test drug administration; 8. Participants voluntarily joined the study and signed informed consent, with good compliance and cooperation with follow-up.

Exclusion Criteria:

- 1. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction; 2. Patients with urinary protein positive (urinary protein detection 2+ or more, or 24-hour urine protein quantification> 1.0g); 3. Patients with hypertension who cannot be reduced to normal range with antihypertensive medication (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg) 4. Concurrent active cancer that requires non-surgical treatment (eg chemotherapy, radiotherapy, adjuvant therapy) 5. Previously suffered severe cardiovascular disease: myocardial ischemia or myocardial infarction of grade Ⅱ or above, poorly controlled arrhythmia (including QTc interval ≥450 ms for men, ≥470 ms for women); according to NYHA standards, grade Ⅲ ～ Ⅳ Cardiac insufficiency, or color Doppler ultrasound examination of the left ventricular ejection fraction (LVEF) <50%; 6. For previous symptoms of cerebral hemorrhage of grade 2 or higher, bleeding in other parts of grade ≥CTCAE grade 3 occurred within 4 weeks before the first use of the study drug; 7. Abnormal blood coagulation function (International Normalized Ratio of Prothrombin Time (INR)> 1.5 ULN or Prothrombin Time (PT)> ULN + 4 seconds or APTT> 1.5 ULN), with bleeding tendency 8. Patients who are receiving thrombolytic or anticoagulant therapy and treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; small-dose prophylaxis is allowed for preventive purposes provided that INR is ≤1.5 Warfarin (1mg orally, once daily) or low-dose aspirin (between 80mg and 100mg daily); 9. Arterial / venous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism, occurring within 6 months before the first medication; 10. Severe or non-healing wounds, ulcers or fractures or abdominal fistulas, gastrointestinal perforations, abdominal abscesses, major medical history of open biopsy or significant trauma within 28 days prior to administration except for craniotomy and tumor removal 11. The researcher judges other situations that may affect the progress of the clinical study and the determination of the research results, and considers them unsuitable for inclusion.

12. Pregnant or lactating women; 13. Have previously used other anti-angiogenic drugs or preparations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | up to 1 year
  Proportion of progression-free survival up to 6 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 1 year
  Refers to the date from the random date to the first occurrence of disease progression or death from any cause, whichever occurs first.
Overall survival (OS) | up to 1 year
  Means from random date to the date of death for any reason
Objective response rate (ORR) | up to 1 year
  Refers to the proportion of patients whose tumors have shrunk to a certain level and maintained for a certain period of time, including cases of CR and PR. The solid tumor remission assessment standard (RECIST 1.1) was used to evaluate the objective tumor remission.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wu, archiater, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China